CLINICAL TRIAL: NCT07023770
Title: Rehabilitation Program Dedicated to Post-stroke Lateropulsion Including Exoskeleton Assisted Exercises
Acronym: EXOLAT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Fondation pour la recherche sur les AVC (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 38RC24.0254; 2024-A01586-41 (Other: Grenoble University Hospital)
Record Dates: First submitted 2025-04-22; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Stroke, Ischemic
Keywords: lateropulsion; exoskeleton; rehabilitation program
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Multiple baseline designs of a " single case experimental design " applied in 3 participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- program week 2-3-4 (Experimental): For the participant included in this arm, the intervention will take place during weeks 2-3-4 (5 times per week 30-min sessions with specific physiotherapy targeting lateropulsion including exercices in exoskeleton + 5 times per week conventional physiotherapy). During weeks 1, 5, 6, 7 & 8, 30-min sessions of conventional physiotherapy will take place 10 times per week. The rest of the rehabilitation (speech therapy, neuropsychology, occupational therapy) will be provided as usual.
  Interventions: Behavioral: specific lateropulsion rehabilitation program (exoskeleton + specific physiotherapy orientation rehabilitation); Behavioral: Conventional physiotherapy without without exercises dedicated to lateropulsion or verticality representation alleviation
- program week 3-4-5 (Experimental): For the participant included in this arm, the intervention will take place during weeks 3-4-5 (5 times per week 30-min sessions with specific physiotherapy targeting lateropulsion including exercices in exoskeleton + 5 times per week conventional physiotherapy). During weeks 1, 2, 6, 7 & 8, 30-min sessions of conventional physiotherapy will take place 10 times per week. The rest of the rehabilitation (speech therapy, neuropsychology, occupational therapy) will be provided as usual.
  Interventions: Behavioral: specific lateropulsion rehabilitation program (exoskeleton + specific physiotherapy orientation rehabilitation); Behavioral: Conventional physiotherapy without without exercises dedicated to lateropulsion or verticality representation alleviation
- program week 4-5-6 (Experimental): For the participant included in this arm, the intervention will take place during weeks 4-5-6 (5 times per week 30-min sessions with specific physiotherapy targeting lateropulsion including exercices in exoskeleton + 5 times per week conventional physiotherapy). During weeks 1, 2, 3, 7 & 8, 30-min sessions of conventional physiotherapy will take place 10 times per week. The rest of the rehabilitation (speech therapy, neuropsychology, occupational therapy) will be provided as usual.
  Interventions: Behavioral: specific lateropulsion rehabilitation program (exoskeleton + specific physiotherapy orientation rehabilitation); Behavioral: Conventional physiotherapy without without exercises dedicated to lateropulsion or verticality representation alleviation

INTERVENTIONS:
Behavioral: specific lateropulsion rehabilitation program (exoskeleton + specific physiotherapy orientation rehabilitation) — 5 times a week during 30 minutes sessions = 15 Physiotherapy sessions, focused on the active vertical body orientation in the frontal plane and comprising exoskeleton-assisted balance and gait exercises.
  + 5 times a week during 30 minutes sessions = 15 conventional physiotherapy without exercises dedicated to lateropulsion or verticality representation alleviation The intervention description is more extensive in the study description section
Behavioral: Conventional physiotherapy without without exercises dedicated to lateropulsion or verticality representation alleviation — 10 times a week, during 30-minutes

SUMMARY:
Lateropulsion is a deficit in the body orientation with respect to the vertical in the coronal plane, defined by the presence of one of the three signs: lateral body tilt, active pushing from the sound limbs, and resistance to passive corrections. The lateral body tilt is the cardinal sign, the frequency of the 2 other signs increasing with lateropulsion severity (most dramatic forms called pusher syndrome in the past). Lateropulsion is frequent after stroke, and represents the main factor underpinning balance and gait disorders at the subacute phase. After hemisphere stroke lateropulsion is caused by a bias in the internal model of the verticality in the frontal plane, individuals unconsciously aligning their body posture on a tilted verticality representation. Pilot studies suggested the possibility to recalibrate the internal model of verticality, biased by stroke, and to improve individuals' uprightness. The investigators expect that a specific rehabilitation program combining technics devoted to lateropulsion, and comprising exoskeleton (Atalante) assisted balance exercises could help recalibrate the internal model of verticality and alleviate lateropulsion. The primary objective is to test the hypothesis that a 3-week specific lateropulsion rehabilitation program (15 sessions of 30 minutes including exoskeleton and a rehabilitation focused on the vertical body orientation in the frontal plane) improves the visual vertical (VV), the most used test to assess verticality perception.

DETAILED DESCRIPTION:
BACKGROUND To our knowledge, no study has ever assessed the effects of a rehabilitation program specifically devoted to lateropulsion. The investigators expect that such a specific program combining different technics selected on the basis of theoretical rationale, experimental evidence in healthy subjects, or phase I-II randomized clinical studies, and supposed to improve verticality representation or alleviate lateropulsion could improve verticality representation and alleviate lateropulsion. The investigators hypothesize that individuals with moderate to severe lateropulsion after hemisphere stroke could benefit from such a specific lateropulsion rehabilitation program.

OBJECTIVES The primary objective is to test the hypothesis that, in individuals with a first ischemic right hemisphere stroke showing a moderate to severe lateropulsion due to a biased internal model of verticality, a 3-week intensive specific and intensive lateropulsion rehabilitation program (15 physiotherapy sessions of 30 minutes including exoskeleton-assisted lateral balance exercises) improves the visual perception of the verticality as assessed by the Visual Vertical (VV) orientation. This outcome has been selected because it may be repeatedly assessed, which is necessary in a Small-N design Study.

The secondary objectives are to:

* Test the hypothesis that the specific and intensive lateropulsion rehabilitation program also modulates the postural perception of the vertical (PV). This transmodal modulation of verticality perception involving both VV and PV would mean that the internal model of verticality has been recalibrated. This would have a clinical and scientific significance going far beyond a simple change in verticality perception
* Test the hypothesis that the specific and intensive lateropulsion rehabilitation program alleviates lateropulsion;
* Test the hypothesis that the specific and intensive lateropulsion rehabilitation program improves balance and gait abilities without any effect on the motricity of the paretic upper limb;
* Evaluate the participants' perception at the end of this specific rehabilitation program.

HYPOTHESES Considering the main objective, the investigators hypothesize that the specific and intensive lateropulsion rehabilitation program will improve VV orientation of at least 2°, constituting a real change in VV perception.

STUDY DESIGN The study is a monocentric Small-n design study. The experimental plan is a multiple baseline design. This design applies for intervention with slow/delayed changes and no expected washout. Three participants will be included after about the same time post stroke (subacute phase). The VV will be measured daily (except on weekends) for each participant (i.e. 5 VV per week ), and the generalization and control measures measured once each week. All participants will follow a conventional rehabilitation program until they start the intervention.

One participant will start the intervention period 2 weeks after enrolment. Another will start at 3 weeks after enrolment and the last one will start at 3 weeks after enrolment. All participants will be assessed repetitively on the target variables. The sequential introduction of the intervention in 3 participants will allow the visualization of lack of retest effect and of progress unrelated to intervention in the individuals not having the intervention yet.

INTERVENTION

During the baseline and after the 3-week intervention, individuals will follow the conventional rehabilitation program including :

* 2 sessions per day of 30-minutes of "conventional" physiotherapy 5 days a week without exercises specifically devoted to the control of body orientation in frontal plane, or verticality representation
* 1 session of 30-min of occupational therapy 5 days a week
* speech therapy and neuropsychology if necessary.

During the 3-week intervention, individuals will have:

* 1 session per day of 30-min of physiotherapy specifically focused on the body orientation with respect to gravity in the frontal plane, including exoskeleton-assisted balance and gait exercises 3 times a week, 5 days a week,
* 1 session per day of 30-min conventional physiotherapy 5 days a week
* 1 session of 30-min of occupational therapy 5 days a week
* speech therapy and neuropsychology if necessary. So, the intervention phase lasts 3 weeks, and consists in 15 physiotherapy sessions, focused on the active vertical body orientation in the frontal plane and comprising exoskeleton-assisted balance and gait exercises. Participants have the same dose of rehabilitation in each phase (baseline, during intervention and after intervention), which only differ in the nature of the rehabilitation.

During the specific rehabilitation program, the frame of exercises with the Atalante® exoskeleton comprises verticalization: work in standing position, stepping, walking in different directions including backward, with the help of a mirror or without visual information (eyes closed). Some exercises in the exoskeleton will also be performed when the participant is laterally tilted (in a static position, during active functional tasks, eyes open and closed).

The specific physiotherapy rehabilitation targeting lateropulsion will include: verticality awareness, exercises in front of a mirror to facilitate the awareness of body tilt (or with a video record), posturography with biofeedback, trunk inclination, reaching tasks in sitting and standing position, walking with body-weight support, orientation tasks during sensorial ponderation (eyes open/closed, foam or firm surface, cervical extension...) The investigators chose not to include brain stimulation in this program.

PARTICIPANTS Three patients will be included. The study will be explained to eligible individuals who will be free to participate or not. An informed consent form will then be signed by each participant.

To meet the scientific standards of SCEDs, one required design criteria is to include at least three attempts to demonstrate an intervention effect (i.e. 3 participants in our case). The sequential introduction of the intervention in 3 participants will allow the visualization of effect of the intervention on the VV.

RELEVANCE Regaining independent balance and mobility is a major goal in post-stroke rehabilitation. While lateropulsion due to a biased internal model of verticality is one of the most important detrimental factors affecting balance and gait at the post-stroke subacute phase, no specific lateropulsion rehabilitation program has ever been scientifically validated with a high level of evidence. This study will focus on individuals with moderate to severe lateropulsion caused by a biased internal model of verticality due to a right hemisphere stroke which are known to have lesser recovery and longer hospital length of stay. A specific and intensive lateropulsion rehabilitation program dedicated to the active vertical body orientation in the frontal plan could speed up the mobility recovery and shorten the hospitalization period.

ELIGIBILITY:
Inclusion Criteria:

* Right hemispheric first and unique ischemic stroke between 2 weeks and 6 months old (subacute phase) ;
* Presence of lateropulsion, assessed by the Scale for Contraversive Pushing (2 ≤ SCP < 5)
* Presence of contralesional VV bias (VV > 4°)
* Right handedness defined by a Edinburgh score ≥0,39
* Being hospitalized in a Physical Medicine and Neurological Rehabilitation (PMR) facility.
* Have given a written and informed consent

Exclusion Criteria:

* Medical instability making evaluation impossible,
* Comprehension or cognitive or behavioral disorders, or depressive symptoms that compromise participation in the program
* Postural disorders or body geometry disorders that interfere with balance for a reason that is independant of the stroke
* Morphological contraindications to the use of the Atalante® robot (segment length or joint ranges; height <155cm; weight >100kg),
* Severe spasticity (>3 on the modified Ashworth scale) in the adductors, quadriceps, hamstrings and triceps surae
* Presence of a pressure sore at the areas of contact with the Atalante® robot,
* History of osteoporotic fractures.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2025-06-20 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Visual Vertical (VV) Orientation | Daily, from enrollment to the end of treatment at 8 weeks
  VV consists in testing the direction of a visual line, perceived as vertical by participants, in complete darkness. VV will be tested by a well-validated apparatus and paradigm (Pérennou et al Brain 2008 ; Piscicelli & Pérennou 2017). VV orientation will be the average orientation (in degree) of the 10 trials performed. Higher score means a worse outcome, indicating the magnitude of the bias in verticality perception.

SECONDARY OUTCOMES:
Postural Vertical (PV) orientation and uncertainty | Once a week from enrollment to the end of program at 8 weeks
  PV consists in testing the whole body orientation in sitting, perceived as vertical by participants, in complete darkness. PV will be tested by a well-validated apparatus and paradigm (Pérennou et al Brain 2008). PV orientation will be the average orientation (in degree) of the 10 trials performed ; PV uncertainty is the standard deviation of the 10 trials performed in degrees. Higher scores mean worse outcomes, indicating the magnitude of the bias in verticality perception
Lateropulsion severity assessed by SCALA | once a week from enrollment to the end of treatment at 8 weeks
  The SCAle for LAteropulsion (SCALA) scores range from 0 (no lateropulsion) to 50 (severe lateropulsion with pushing); higher scores mean a worse outcome
Lateropulsion severity assessed by SCP | once a week from enrollment to the end of treatment at 8 weeks
  The SCP (= clinical Scale for Contraversive Pusching, Karnath et al. (2000)) scores range from 0 (no lateropulsion) to 6 (severe lateropulsion with pushing); higher scores mean a worse outcome
Visual Vertical Uncertainty | Daily, from enrollment to the end of treatment at 8 weeks
  VV consists of testing the direction of a visual line, perceived as vertical by particpants, in complete darkness. VV will be tested by a well-validated apparatus and paradigm (Pérennou et al Brain 2008 ; Piscicelli & Pérennou 2017). VV uncertainty will be the standard deviation of the 10 trials performed in degrees. Higher score means a worse outcome.
specific post-effect of one exoskeleton session on visual vertical | once a week during the 3 lateropulsion program weeks
  orientation of VV in degrees, a higher score indicate a higher verticality perception biais.
  15 minutes max after exoskeleton session.
Lower limb motricity assessed by "Fugl-Meyer Assessment of Motor Recovery after Stroke" | once a week from enrollment to the end of treatment at 8 weeks
  Motor score of lower extremity ranges from 0 (hemiplegia) 34 points (normal motor performance). A higher score means a better outcome.
Balance assessed by the modified Postural Assessment Scale for Stroke (mPASS) total score | once a week from enrollment to the end of the study at week 8
  The modified Postural Assessment Scale for Stroke patient (m-PASS) scores range from 0 (poorer balance ability) to 50 (excellent balance ability). Higher scores mean a better outcome.
Gait assessed by Modified Fugl-Meyer Gait Assessment total score | once a week from enrollment to the end of the study (week 8)
  Modified Fugl-Meyer Gait Assessment score ranges from 0 (not able to walk) to 6 (walks at a normal speed for his age). Higher score means better outcome (Lindmark 1988).
Functionnal mobility | once a week fron enrollment to the end of the study (week 8)
  Time in seconds at the Time up and go test (TUG). Higher time means worse outcome.
Upper limb motricity assessed by "Fugl-Meyer Assessment of Motor Recovery after Stroke" | once a week from enrollment to the end of the treatment (week 8)
  Motor score of upper extremity ranges from 0 (hemiplegia) to 66 points (normal motor performance). A higher score means a better outcome.
Positions (on both anterior and lateral axes) of the center of pression in the exoskeleton while lateraly inclined | During lateropulsion program, Day 1 and Day 5 of the first week, Day 5 of the second week and Day 5 of the third week.
  Measured in the exoskeleton in millimeters. Higher score indicates an asymmetric weight beiring.
Patient reported discomfort experienced during exoskeleton sessions | Once, on day 5 of the third week of the specific and intensive lateropulsion rehabilitation program including exercices in the exoskeleton
  Recorded on a visual analog scale (0-10; lower values better) and a semi-structured interview
Patient reported satisfaction of exoskeleton sessions | Once, on day 5 of the third week of the specific and intensive lateropulsion rehabilitation program including exercices in the exoskeleton
  Recorded on a visual analog scale (0-10; higher values better) and a semi-structured interview
feasibility and satisfaction of the lateropulsion program perceived by physiotherapist | Once, on day 5 of the third week of the specific and intensive lateropulsion rehabilitation program including exercices in the exoskeleton
  physiotherapist point of view, recorded with a semi structured interview and visual analog scales for feasibility and satisfaction ranging from 0 to 10, with higher scores indicating better outcomes
specific effect of exoskeleton practice on positions (on both anterior and lateral axes) of the center of pression in the exoskeleton while lateraly inclined | During lateropulsion program, before and after a training session, on Day 1 and Day 5 of the first week, Day 5 of the second week and Day 5 of the third week.
  Measured in the exoskeleton in millimeters. Higher score indicates an asymmetric weight beiring.

CONTACTS AND LOCATIONS:
Overall Officials: Dominic Pérennou, MD, PhD, Pr, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - Grenoble University Hospital, Échirolles
  - Grenoble University Hospital, Grenoble

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data that support the findings of this study will be available from the principal investigator (Pr Dominic Pérennou), upon reasonable request, only for authorized research. Their use is subjected to an agreement with the promotor (CHU Grenoble) and the principal investigator of the EXOLAT study
Supporting Information: CSR
Time Frame: After seminal publication of the results
Access Criteria: Anonymized data that support the findings of this study will be available from the principal investigator (Pr Dominic Pérennou), upon reasonable request, only for authorized research. Their use is subjected to an agreement with the promotor (CHU Grenoble) and the principal investigator of the EXOLAT study

REFERENCES:
- [Background] Yun N, Joo MC, Kim SC, Kim MS. Robot-assisted gait training effectively improved lateropulsion in subacute stroke patients: a single-blinded randomized controlled trial. Eur J Phys Rehabil Med. 2018 Dec;54(6):827-836. doi: 10.23736/S1973-9087.18.05077-3. Epub 2018 Dec 3. PMID 30507899
- [Background] Winstein CJ, Stein J, Arena R, Bates B, Cherney LR, Cramer SC, Deruyter F, Eng JJ, Fisher B, Harvey RL, Lang CE, MacKay-Lyons M, Ottenbacher KJ, Pugh S, Reeves MJ, Richards LG, Stiers W, Zorowitz RD; American Heart Association Stroke Council, Council on Cardiovascular and Stroke Nursing, Council on Clinical Cardiology, and Council on Quality of Care and Outcomes Research. Guidelines for Adult Stroke Rehabilitation and Recovery: A Guideline for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2016 Jun;47(6):e98-e169. doi: 10.1161/STR.0000000000000098. Epub 2016 May 4. PMID 27145936
- [Background] Piscicelli C, Perennou D. Visual verticality perception after stroke: A systematic review of methodological approaches and suggestions for standardization. Ann Phys Rehabil Med. 2017 Jun;60(3):208-216. doi: 10.1016/j.rehab.2016.02.004. Epub 2016 Apr 11. PMID 27079584
- [Background] Perennou DA, Mazibrada G, Chauvineau V, Greenwood R, Rothwell J, Gresty MA, Bronstein AM. Lateropulsion, pushing and verticality perception in hemisphere stroke: a causal relationship? Brain. 2008 Sep;131(Pt 9):2401-13. doi: 10.1093/brain/awn170. Epub 2008 Aug 4. PMID 18678565
- [Background] Perennou DA, Amblard B, Leblond C, Pelissier J. Biased postural vertical in humans with hemispheric cerebral lesions. Neurosci Lett. 1998 Aug 14;252(2):75-8. doi: 10.1016/s0304-3940(98)00501-1. PMID 9756325
- [Background] Paci M, Macchioni G, Ferrarello F. Treatment approaches for pusher behaviour: a scoping review. Top Stroke Rehabil. 2023 Mar;30(2):119-136. doi: 10.1080/10749357.2021.2016098. Epub 2022 Feb 14. PMID 35156566
- [Background] Odin A, Faletto-Passy D, Assaban F, Perennou D. Modulating the internal model of verticality by virtual reality and body-weight support walking: A pilot study. Ann Phys Rehabil Med. 2018 Sep;61(5):292-299. doi: 10.1016/j.rehab.2018.07.003. Epub 2018 Jul 19. PMID 30031891
- [Background] Nolan J, Jacques A, Godecke E, Abe H, Babyar S, Bergmann J, Birnbaum M, Dai S, Danells C, Edwards TG, Gandolfi M, Jahn K, Koter R, Mansfield A, Nakamura J, Pardo V, Perennou D, Piscicelli C, Punt D, Romick-Sheldon D, Saeys W, Smania N, Vaes N, Whitt AL, Singer B. Clinical practice recommendations for management of lateropulsion after stroke determined by a Delphi expert panel. Clin Rehabil. 2023 Nov;37(11):1559-1574. doi: 10.1177/02692155231172012. Epub 2023 Apr 26. PMID 37122265
- [Background] Louie DR, Mortenson WB, Durocher M, Schneeberg A, Teasell R, Yao J, Eng JJ. Efficacy of an exoskeleton-based physical therapy program for non-ambulatory patients during subacute stroke rehabilitation: a randomized controlled trial. J Neuroeng Rehabil. 2021 Oct 10;18(1):149. doi: 10.1186/s12984-021-00942-z. PMID 34629104
- [Background] Lewis J, Heinemann T, Jacques A, Chan K, Harper KJ, Nolan J. Lateropulsion is a predictor of falls during inpatient stroke rehabilitation. Ann Phys Rehabil Med. 2024 Mar;67(2):101814. doi: 10.1016/j.rehab.2023.101814. Epub 2024 Mar 20. No abstract available. PMID 38513306
- [Background] Krewer C, Riess K, Bergmann J, Muller F, Jahn K, Koenig E. Immediate effectiveness of single-session therapeutic interventions in pusher behaviour. Gait Posture. 2013 Feb;37(2):246-50. doi: 10.1016/j.gaitpost.2012.07.014. Epub 2012 Aug 11. PMID 22889929
- [Background] Hsu TH, Tsai CL, Chi JY, Hsu CY, Lin YN. Effect of wearable exoskeleton on post-stroke gait: A systematic review and meta-analysis. Ann Phys Rehabil Med. 2023 Feb;66(1):101674. doi: 10.1016/j.rehab.2022.101674. Epub 2022 Nov 30. PMID 35525427
- [Background] Fukata K, Amimoto K, Inoue M, Shida K, Kurosawa S, Inoue M, Fujino Y, Makita S, Takahashi H. Effects of performing a lateral-reaching exercise while seated on a tilted surface for severe post-stroke pusher behavior: A case series. Top Stroke Rehabil. 2021 Dec;28(8):606-613. doi: 10.1080/10749357.2020.1861718. Epub 2020 Dec 20. PMID 33345722
- [Background] Dieterich M, Brandt T. Wallenberg's syndrome: lateropulsion, cyclorotation, and subjective visual vertical in thirty-six patients. Ann Neurol. 1992 Apr;31(4):399-408. doi: 10.1002/ana.410310409. PMID 1586141
- [Background] Danells CJ, Black SE, Gladstone DJ, McIlroy WE. Poststroke "pushing": natural history and relationship to motor and functional recovery. Stroke. 2004 Dec;35(12):2873-8. doi: 10.1161/01.STR.0000147724.83468.18. Epub 2004 Nov 4. PMID 15528459
- [Background] Dai S, Piscicelli C, Clarac E, Baciu M, Hommel M, Perennou D. Balance, Lateropulsion, and Gait Disorders in Subacute Stroke. Neurology. 2021 Apr 27;96(17):e2147-e2159. doi: 10.1212/WNL.0000000000011152. Epub 2020 Nov 11. PMID 33177223
- [Background] Dai S, Lemaire C, Piscicelli C, Perennou D. Lateropulsion Prevalence After Stroke: A Systematic Review and Meta-analysis. Neurology. 2022 Apr 12;98(15):e1574-e1584. doi: 10.1212/WNL.0000000000200010. Epub 2022 Feb 21. PMID 35190465
- [Background] Calabro RS, Sorrentino G, Cassio A, Mazzoli D, Andrenelli E, Bizzarini E, Campanini I, Carmignano SM, Cerulli S, Chisari C, Colombo V, Dalise S, Fundaro C, Gazzotti V, Mazzoleni D, Mazzucchelli M, Melegari C, Merlo A, Stampacchia G, Boldrini P, Mazzoleni S, Posteraro F, Benanti P, Castelli E, Draicchio F, Falabella V, Galeri S, Gimigliano F, Grigioni M, Mazzon S, Molteni F, Morone G, Petrarca M, Picelli A, Senatore M, Turchetti G, Bonaiuti D; Italian Consensus Conference on Robotics in Neurorehabilitation (CICERONE). Robotic-assisted gait rehabilitation following stroke: a systematic review of current guidelines and practical clinical recommendations. Eur J Phys Rehabil Med. 2021 Jun;57(3):460-471. doi: 10.23736/S1973-9087.21.06887-8. Epub 2021 May 5. PMID 33947828
- [Background] Brandt T, Dieterich M, Danek A. Vestibular cortex lesions affect the perception of verticality. Ann Neurol. 1994 Apr;35(4):403-12. doi: 10.1002/ana.410350406. PMID 8154866
- [Background] Bergmann J, Krewer C, Jahn K, Muller F. Robot-assisted gait training to reduce pusher behavior: A randomized controlled trial. Neurology. 2018 Oct 2;91(14):e1319-e1327. doi: 10.1212/WNL.0000000000006276. Epub 2018 Aug 31. PMID 30171076
- [Background] Barra J, Marquer A, Joassin R, Reymond C, Metge L, Chauvineau V, Perennou D. Humans use internal models to construct and update a sense of verticality. Brain. 2010 Dec;133(Pt 12):3552-63. doi: 10.1093/brain/awq311. Epub 2010 Nov 19. PMID 21097492
- [Background] Baier B, Suchan J, Karnath HO, Dieterich M. Neural correlates of disturbed perception of verticality. Neurology. 2012 Mar 6;78(10):728-35. doi: 10.1212/WNL.0b013e318248e544. Epub 2012 Feb 22. PMID 22357719
- [Background] Baggio JA, Mazin SS, Alessio-Alves FF, Barros CG, Carneiro AA, Leite JP, Pontes-Neto OM, Santos-Pontelli TE. Verticality Perceptions Associate with Postural Control and Functionality in Stroke Patients. PLoS One. 2016 Mar 8;11(3):e0150754. doi: 10.1371/journal.pone.0150754. eCollection 2016. PMID 26954679
- [Background] Babyar SR, Peterson MG, Reding M. Time to recovery from lateropulsion dependent on key stroke deficits: a retrospective analysis. Neurorehabil Neural Repair. 2015 Mar-Apr;29(3):207-13. doi: 10.1177/1545968314541330. Epub 2014 Jul 8. PMID 25009223
- [Background] An CM, Ko MH, Kim DH, Kim GW. Effect of postural training using a whole-body tilt apparatus in subacute stroke patients with lateropulsion: A single-blinded randomized controlled trial. Ann Phys Rehabil Med. 2021 Mar;64(2):101393. doi: 10.1016/j.rehab.2020.05.001. Epub 2020 Oct 14. PMID 32450273
- [Background] Abe H, Kondo T, Oouchida Y, Suzukamo Y, Fujiwara S, Izumi S. Prevalence and length of recovery of pusher syndrome based on cerebral hemispheric lesion side in patients with acute stroke. Stroke. 2012 Jun;43(6):1654-6. doi: 10.1161/STROKEAHA.111.638379. Epub 2012 Mar 1. PMID 22382159